CLINICAL TRIAL: NCT05981755
Title: Breathing Rescue for SUDEP Prevention (BreatheS)
Brief Title: Breathing Rescue for SUDEP Prevention
Acronym: BreatheS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nuria Lacuey Lecumberri, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-20-1228; R01NS133743 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-08-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Brain Mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Breathing tasks and Brain mapping with stimulation (Experimental)
  Interventions: Other: Breathing tasks; Device: Brain mapping with stimulation

INTERVENTIONS:
Other: Breathing tasks — Breathing tasks include normal breathing through nose or mouth, breathing while resting wakefully, increase and decrease in breathing rate, and breath counting.
Device: Brain mapping with stimulation — Electrical stimulation will be used to find specific areas of the brain involved in breathing function. Stimulation will be applied using a Nihon Kohden MEE-1000A neural function measuring system with the MS-120BK extension unit for brain stimulation.

SUMMARY:
The purpose of this study is to precisely delineate human brain networks that modulate respiration and identify specific brain areas and stimulation techniques that can be used to prevent seizure-induced breathing failure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of intractable focal epilepsy
* admitted to the Epilepsy Monitoring Unit (EMU) at Memorial Hermann-Texas Medical Center for intracranial subdural strips, grids, or depth electrode placement study (invasive video-EEG)

Exclusion Criteria:

* respiratory, cardiac or cerebrovascular disease
* pregnancy
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of breathing node size as assessed by electroencephalogram (EEG) signal | baseline (before breathing task), at the time of the breathing task (about 8 minutes after start of baseline)
Change in presence of breathing nodes as assessed by EEG signal | Baseline (before breathing task), at the time of the breathing task(about 8 minutes after start of baseline)
Changes in thoracoabdominal circumference during stimulation as assessed by thoracoabdominal belts, | Baseline, during the stimulation session (at least 2 hours after baseline)
  Lower and higher frequencies up to 50 Hertz(Hz), current of 1-10 milli ampere (mA), pulse durations of 0.2 milli second (msec) and stimulation periods of 10 to 40 seconds will be used.
Changes airflow during stimulation as assessed by the nasal/oral pressure transducer [BiNAPS] | Baseline, during the stimulation session (at least 2 hours after baseline)
  Lower and higher frequencies up to 50Hz, current of 1-10mA, pulse durations of 0.2 msec and stimulation periods of 10 to 40 seconds will be used.
Change in Saturation of peripheral oxygen (SpO2) during stimulation as assessed by the pulse oximetry | Baseline, during the stimulation session (at least 2 hours after baseline)
  Lower and higher frequencies up to 50Hz, current of 1-10mA, pulse durations of 0.2 msec and stimulation periods of 10 to 40 seconds will be used.
Change in end tidal carbon dioxide (CO2) during stimulation | Baseline, during the stimulation session (at least 2 hours after baseline)
  Lower and higher frequencies up to 50Hz, current of 1-10mA, pulse durations of 0.2 msec and stimulation periods of 10 to 40 seconds will be used.

SECONDARY OUTCOMES:
Quantification of the breathing changes as assessed by the change in breathing rate | baseline (before stimulation), at the time of stimulation (about 8 minutes after start of baseline)
  Breathing rate is the number of breaths taken per minute. Breathing changes will be visually identified live during stimulation sessions using thoraco-abdominal plethysmography and pressure transducer signal (nasal/oral airflow).
Quantification of the breathing changes as assessed by the change in breathing depth | baseline (before stimulation), at the time of stimulation (about 8 minutes after start of baseline)
  Breathing depth, or tidal volume (TV), is the amount of air that normally enters the lungs during quiet breathing. Breathing changes will be visually identified live during stimulation sessions using thoraco-abdominal plethysmography and pressure transducer signal (nasal/oral airflow).
Quantification of the breathing changes as assessed by the change in breathing minute ventilation (MV) | baseline (before stimulation), at the time of stimulation (about 8 minutes after start of baseline)
  Minute ventilation, also known as total ventilation, is a measurement of the amount of air that enters the lungs per minute. It is the product of respiratory rate and tidal volume. Breathing changes will be visually identified live during stimulation sessions using thoraco-abdominal plethysmography and pressure transducer signal (nasal/oral airflow).

CONTACTS AND LOCATIONS:
Overall Officials: Nuria L Lecumberri, MD,PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No